CLINICAL TRIAL: NCT00716560
Title: Nausea and Vomiting In Patients Receiving Consecutive Days of Cisplatin
Status: Terminated | Type: Observational
Why Stopped: Administratively terminated.
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Other Study IDs: 05C.202; 2004-101 (Other: CCRRC); 0402005015 (Other Grant/Funding Number: Merck & Co, Inc.); JT 1069 (Other: JeffTrial Number)
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Melanoma; Nausea
MeSH Terms: conditions — Melanoma; Nausea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Metastatic melanoma treatment with Dartmouth regimen

SUMMARY:
The purpose of this study is to observe the incidence of nausea with systemic chemotherapy that includes consecutive days (more than one day)of cisplatin medication.

DETAILED DESCRIPTION:
Questionnaires are completed on week of chemotherapy treatment referred to as Dartmouth regimen.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis metastatic melanoma
* 18 years and older
* undergoing chemotherapy with Dartmouth regimen
* medically stable to receive chemotherapy per physical and clinical laboratory tests

Exclusion Criteria:

* No medical conditions that interfere with assessment of nausea and vomiting during chemotherapy
* No cognitive disorder that impairs symptom assessment
* No other investigational agent
* Inability to swallow medications for nausea and vomiting
* No gastric outlet obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University practice patients with metastatic melanoma
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2005-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Determine incidence of nausea when receiving Dartmouth regimen chemotherapy for metastatic melanoma | Week of treatment

SECONDARY OUTCOMES:
Assess the impact of systemic chemotherapy with Dartmouth regimen on quality of life of patients | week of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Takami Sato, M.D.,Ph.D., Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University — http://www.KimmelCancerCenter.org